CLINICAL TRIAL: NCT03274466
Title: Post-market, Randomized, Open-Label, Multicenter, Study to Evaluate the Effectiveness of Closed Incision Negative Pressure Therapy Versus Standard of Care Dressings in Reducing Surgical Site Complications in Subjects With Revision of a Failed Total Knee Arthroplasty (PROMISES)
Brief Title: Closed Incision Negative Pressure Therapy Versus Standard of Care Surgical Dressing in Revision Total Knee Arthroplasty
Acronym: PROMISES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KCI USA, Inc (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCI.PREVENA.2017.01
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Results first posted 2021-02-10 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Surgical Wound; Revision Total Knee Arthroplasty; Wounds and Injuries; Joint Disease; Musculoskeletal Disease; Prosthesis-Related Infections; Infection; Postoperative Complications; Pathologic Processes
MeSH Terms: conditions — Surgical Wound; Wounds and Injuries; Joint Diseases; Musculoskeletal Diseases; Prosthesis-Related Infections; Infections; Postoperative Complications; Pathologic Processes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Closed Incision Negative Pressure Therapy (ciNPT) (Experimental): Prevena Peel & Place or Prevena Plus Customizable Dressing and ActiVAC Therapy Unit or Prevena Plus Therapy Unit
  Interventions: Device: Closed Incision Negative Pressure Therapy (ciNPT)
- Standard of Care Dressing (Active Comparator): Silver impregnated dressing
  Interventions: Device: Standard of Care Dressing

INTERVENTIONS:
Device: Closed Incision Negative Pressure Therapy (ciNPT) — Closed Incision Negative Pressure Therapy applied through a foam bolster with a wicking interface fabric that includes 0.019% ionic silver at 125 mmHg of negative pressure for 5-7 days.
  Other Names: Prevena Peel & Place; Prevena Plus Customizable; ActiV.A.C. Therapy Unit; Prevena Plus 125 Therapy Unit
  Arms: Closed Incision Negative Pressure Therapy (ciNPT)
Device: Standard of Care Dressing — A standard silver-impregnated dressing applied to a closed surgical incision for 5-7 days post-operatively.
  Other Names: Silver-impregnated dressing, Aquacel Ag Surgical or other equivalent
  Arms: Standard of Care Dressing

SUMMARY:
This study evaluates surgical site complications in subjects undergoing revision of a total knee arthroplasty when closed incision negative pressure therapy is used to manage the closed incision, as compared to a standard of care dressing.

ELIGIBILITY:
Pre-operative Inclusion Criteria:

The subject:

* is at least 22 years of age on the date of informed consent
* is able to provide their own informed consent
* requires a TKA revision defined as one of the following:

  1. a one-stage aseptic revision procedure
  2. a one-stage septic exchange procedure (requiring removal of all hardware) for acute postoperative infection
  3. removal of cement spacer and re-implantation procedure
  4. open reduction and internal fixation of peri-prosthetic fractures
* has one or more of the following:

  1. a body mass index (BMI) greater than 35 kg/m2
  2. a requirement for the use of blood thinners other than acetylsalicylic acid (ASA) after surgery
  3. history of or current peripheral vascular disease
  4. the presence of lymphedema in the operative limb
  5. insulin-dependent diabetes mellitus
  6. current tobacco use or previous history of smoking and quitting within the past 30 days
  7. a history of prior infection of the operative site
  8. current use of immunomodulators or steroids
  9. current or history of cancer or hematological malignancy (excluding localized skin cancer)
  10. rheumatoid arthritis
  11. current renal failure or dialysis
  12. malnutrition as determined by the investigator
  13. liver disease as determined by the investigator
  14. status post solid organ transplant
  15. HIV
* is willing and able to return for all scheduled study visits
* if female, has a negative urine or serum pregnancy test at screening and day of revision surgery. Women who have had surgical sterilization by a medically accepted method such as tubal ligation, hysterectomy, or oophorectomy or are post-menopausal, defined as not having menstruation for >= 12 months will be excluded from requiring this test.

Intra-operative Inclusion Criteria:

The subject:

* continues to meet all pre-operative inclusion criteria
* has undergone a TKA revision resulting in a closed surgical incision

Pre-operative Exclusion Criteria:

The subject:

* is pregnant or lactating
* will undergo a bilateral TKA within the same operative visit
* will undergo a bilateral TKA in which the first TKA surgery is on the knee selected for study
* will undergo a staged bilateral TKA in which the TKA revision surgery for the knee under study occurs within 30 days of the first TKA procedure
* was previously randomized in this protocol
* has a systemic active infection at the time of revision not including chronic viral infections such as HIV or hepatitis
* has a remote-site skin infection at the time of revision
* was tattooed on the area of the incision within 30 days prior to randomization
* has known sensitivity to the study product components (drape and/or dressing materials in direct contact with the closed incision or skin)
* has known sensitivity to silver
* is currently enrolled in another investigational trial that requires additional interventions
* is planned to be enrolled in another investigational trial that requires additional interventions at any time during the study
* has localized skin cancer around the incision site

Intra-operative Exclusion Criteria:

The subject:

* is found to meet any of the pre-operative exclusion criteria
* has a surgical incision that precludes placement of dressing
* has a TKA revision resulting in a muscle flap
* has a TKA revision resulting in the placement of a spacer
* has an incision drainage and debridement procedure only
* has a surgical incision closed with skin glue

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Higuera, MD, Principal Investigator — The Cleveland Clinic
Locations (17):
- United States (17):
  - Cleveland Clinic, Weston, Florida
  - Emory University Orthopedics & Spine Hospital, Tucker, Georgia
  - LSU Health Science Center, New Orleans, Louisiana
  - University of Missouri Health Care, Columbia, Missouri
  - Northwell Health - SouthSide Hospital, Bay Shore, New York
  - New York University (NYU), New York, New York
  - Hospital for Special Surgery, New York, New York
  - Columbia University Medical Center/New York Presbyterian Hospital, New York, New York
  - Northwell Health - Lenox Hill Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Joint Implant Surgeons, New Albany, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rothman Institute - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Houston Methodist Research Institute, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) | Standard of Care Dressing
Started | 147 | 147
Completed | 124 | 118
Not Completed | 23 | 29
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Protocol Specified Withdrawal | 5 | 11
Not completed — Lost to Follow-up | 5 | 7
Not completed — Subject Non-compliance | 0 | 1
Not completed — Adverse Event | 3 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 3 | 3

BASELINE CHARACTERISTICS:
Population: Randomized Subjects (ITT)
Groups:
- Total: Total of all reporting groups
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) | Standard of Care Dressing | Total
Number analyzed (Participants) | 147 | 147 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.48) | 65.1 (8.51) | 64.9 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 92 | 175
  Male | 64 | 55 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 6 | 20
  Not Hispanic or Latino | 125 | 134 | 259
  Unknown or Not Reported | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 44 | 50 | 94
  White | 91 | 88 | 179
  More than one race | 10 | 8 | 18
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 147 | 147 | 294
Height [Mean (Standard Deviation); unit: centimeters] — centimeters Population: Data missing from 1 subject.
  centimeters
    number analyzed (Participants) | 147 | 146 | 293
    (all) | 169.8 (10.39) | 168.3 (10.58) | 169.1 (10.49)
Weight [Mean (Standard Deviation); unit: kilograms] — kilograms
  kilograms | 100.4 (21.79) | 96.6 (22.08) | 98.5 (21.98)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Data missing for 1 subject.
  kg/m^2
    number analyzed (Participants) | 147 | 146 | 293
    (all) | 34.7 (6.73) | 34.2 (7.18) | 34.5 (6.96)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Surgical Site Complications (SSC)
Description: The subject incidence of Investigator-assessed surgical site complications (SSCs) within 90 days of TKA revision. SSCs include any of the following:
  * Superficial Surgical Site Infection (SSI)
  * Deep SSI
  * Full thickness skin dehiscence
  * Seroma or hematoma requiring drainage or surgery
  * Skin necrosis
  * Continued drainage at the time of dressing removal
Time Frame: within 90 days after TKA revision
Population: Modified Intent-To-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) | Standard of Care Dressing
Number analyzed (Participants) | 125 | 128
Participants | 5 | 21
Statistical Analysis 1: Comparison: Closed Incision Negative Pressure Therapy (ciNPT) vs Standard of Care Dressing; Test type: Superiority — Modified Intent-To-Treat; p = 0.0013, Cochran-Mantel-Haenszel — Threshold for statistical significance: alpha = 0.048; Odds Ratio (OR) = 0.22, 95% CI 2-sided [0.08 to 0.59]

2. Secondary Outcome: Number of Participants With Surgical Site Infection (SSI) (Superficial or Deep)
Description: 90 day subject incidence of any SSI (superficial or deep)
Time Frame: 90 days after TKA revision
Population: Modified Intent-To-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) | Standard of Care Dressing
Number analyzed (Participants) | 125 | 128
Participants | 2 | 6
Statistical Analysis 1: Comparison: Closed Incision Negative Pressure Therapy (ciNPT) vs Standard of Care Dressing; Test type: Superiority — Modified Intent-To-Treat; p = 0.1680, Cochran-Mantel-Haenszel — Threshold for Statistical Significance: alpha = 0.048; Odds Ratio (OR) = 0.33, 95% CI 2-sided [0.07 to 1.70]

3. Secondary Outcome: Number of Participants With Deep Surgical Site Infection
Description: 90 day subject incidence of deep surgical site infection
Time Frame: 90 days after TKA revision
Population: Modified Intent-To-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) | Standard of Care Dressing
Number analyzed (Participants) | 125 | 128
Participants | 1 | 3
Statistical Analysis 1: Comparison: Closed Incision Negative Pressure Therapy (ciNPT) vs Standard of Care Dressing; Test type: Superiority — Modified Intent-To-Treat; p = 0.3386, Cochran-Mantel-Haenszel — Threshold for Statistical Significance: alpha = 0.048; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.04 to 3.39]

4. Other Pre Specified Outcome: Number of Participants With Surgical Site Complication (SSC)
Description: The subject incidence of Investigator-assessed surgical site complications (SSCs) within 90 days of TKA revision. SSCs include any of the the following:
  * Superficial Surgical Site Infection (SSI)
  * Deep SSI
  * Full thickness skin dehiscence
  * Seroma or hematoma requiring drainage or surgery
Time Frame: within 90 days after TKA revision
Population: Intent-To-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) | Standard of Care Dressing
Number analyzed (Participants) | 147 | 147
Participants | 5 | 21
Statistical Analysis 1: Comparison: Closed Incision Negative Pressure Therapy (ciNPT) vs Standard of Care Dressing; Sensitivity analysis of the Primary Endpoint using the Intent-To-Treat population; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel — Threshold for statistical significance: alpha = 0.048; Odds Ratio (OR) = 0.22, 95% CI 2-sided [0.08 to 0.59]

ADVERSE EVENTS:
Time Frame: 104 days
Description: The Safety Population was utilized for reporting purposes. The Safety Population includes all randomized subjects with at least 1 application of study treatment. Subjects that were randomized but did not receive application of study treatment were withdrawn from the study and therefore not included in the Safety Population. Subjects in the Safety Population were counted under the treatment received irrespective of the assigned treatment.
Arm/Group | Closed Incision Negative Pressure Therapy (ciNPT) | Standard of Care Dressing
All-Cause Mortality (participants affected / at risk) | 1/149 | 0/140
Serious Adverse Events (participants affected / at risk) | 17/149 | 23/140
Other Adverse Events (participants affected / at risk) | 24/149 | 24/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed Incision Negative Pressure Therapy (ciNPT) (N=149) | Standard of Care Dressing (N=140)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Clostridium difficile colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Hypertensive Heart Disease (Cardiac disorders) | 1 (1) | 0 (0) — Hypertensive Coronary Disease Death
Fibrosis (General disorders) | 2 (2) | 1 (1)
Swelling (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 2 (2) | 1 (1)
Stitch abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis infective (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Mental status change (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Arthrotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Joint manipulation (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 3 (3)
Wound drainage (Surgical and medical procedures) | 0 (0) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closed Incision Negative Pressure Therapy (ciNPT) (N=149) | Standard of Care Dressing (N=140)
Blister (Injury, poisoning and procedural complications) | 8 (8) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 7 (7)
Wound Drainage (Surgical and medical procedures) | 8 (8) | 12 (13)
Pain (General disorders) | 4 (5) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT03274466/Prot_001.pdf
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT03274466/SAP_000.pdf